CLINICAL TRIAL: NCT03338348
Title: A Phase II Study With a Safety Run-in Phase Evaluating Vosaroxin With Azacitidine in Older Patients With Newly Diagnosed Acute Myeloid Leukemia and Intermediate/Adverse Genetic Risk or Myelodysplastic Syndrome With Excess Blasts-2 (MDS-EB-2) - AMLSG 24-15
Brief Title: Study of Vosaroxin With Azacitidine in Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome With Excess Blasts-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Sunesis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Verena Gaidzik, Prinicipal Investigator, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 24-15
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts-2 (MDS-EB-2)
Keywords: Vosaroxin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — vosaroxin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine + Vosaroxin (Other): Cycle 1-8:
  Azacitidine: 75 mg/m²/d subcutaneously, d 1-7; Vosaroxin: Dose Level 0: 70mg/m², Dose Level -1: 50mg/m², Dose Level -2: 40mg/m², IV over ten minutes, d 1+4 .
  Patients who have completed 8 cycles of azacitidine and vosaroxin are scheduled to maintenance with single agent azacitidine at 75 mg/m²/d on days 1-7 until relapse or progression.
  Interventions: Drug: Vosaroxin; Drug: Azacitidine

INTERVENTIONS:
Drug: Vosaroxin — Cycle 1-8: Dose Level 0: 70mg/m², Dose Level -1: 50mg/m², Dose Level -2: 40mg/m², IV over ten minutes, d 1+4 .
Drug: Azacitidine — Cycle 1-8 Azacitidine: 75 mg/m²/d subcutaneously, d 1-7;
  Maintenance with single agent azacitidine at 75 mg/m²/d on days 1-7 until relapse or progression.

SUMMARY:
The main part of this trial is a phase II study of vosaroxin with azacitidine in older patients with newly diagnosed AML and intermediate or adverse genetic risk or MDS-EB-2. An initial safety run-in phase of the study will be performed administering the study drug vosaroxin with azacitidine in up to 18 patients. After completion of the run-in phase, toxicity and response data will be provided to the external Data and Safety Monitoring Board (DSMB) and the Trial Committee by the Coordinating Investigator. The Trial Committee will decide on the basis of these data and the recommendation of the DSMB on dose modification and the vosaroxin dose for the phase II part of the study, which will include 150 patients in total.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of acute myeloid leukemia (WHO 2016) and intermediate or adverse genetic risk (according to 2017 ELN recommendations); or patients with myelodysplastic syndrome with excess blasts-2 (MDS-EB-2)
2. Patients ≥60 years of age
3. No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis for up to 10 days during the diagnostic screening phase; patients may have received prior therapy for myelodysplastic syndrome different from hypomethylating agents
4. ECOG performance status ≤2
5. Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 3 month after the last dose of vosaroxin)
6. Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
7. Female patients of reproductive age must agree to avoid getting pregnant while on therapy and for 3 months after the last dose of vosaroxin.
8. Women of child-bearing potential including the female partners of the male patients must either commit to continued abstinence from heterosexual intercourse or apply two acceptable methods of birth control (IUD, tubal ligation, or partner's vasectomy). Hormonal contraception is an inadequate method of birth control.
9. Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy (while on therapy and for three months after the last dose of chemotherapy)
10. Willing to adhere to protocol specific requirements
11. Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out

Exclusion Criteria:

1. Known or suspected hypersensitivity to the study drugs and/or any excipients
2. Favorable genetics: t(15;17)(q22;q12), PML-RARA; t(8;21)(q22;q22), RUNX1-RUNX1T1; inv(16)(p13.1q22)/t(16;16)(p13.1;q22), CBFB-MYH11; mutated NPM1 without FLT3-ITD or with FLT3-ITDlow
3. Prior treatment for AML except hydroxyurea
4. Prior treatment for MDS with hypomethylating agents
5. ECOG performance status >2
6. Patients who are not eligible for intensive chemotherapy
7. Inadequate cardiac, hepatic and/or renal function at the Screening Visit defined as:

   * Ejection fraction <40% confirmed by echocardiography
   * Creatinine >1.5x upper normal serum level
   * Total bilirubin, AST or ALT >1.5 upper normal serum level
8. Active central nervous system involvement
9. Any clinically significant, advanced or unstable disease or history of that may interfere with primary or secondary variable evaluations or put the patient at special risk, such as:

   * Myocardial infarction, unstable angina within 3 months before screening
   * Heart failure NYHA III/IV
   * Severe obstructive or restrictive ventilation disorder
   * Uncontrolled infection
10. Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
11. Currently receiving a therapy not permitted during the study, as defined in Section 10.5.4
12. Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
13. Known history of positive test for Hepatitis B surface Antigen (HBsAg) or hepatitis C antibody or history of positive test for Human Immunodeficiency Virus (HIV)
14. Hematological disorder independent of leukemia
15. No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation
16. No consent for biobanking
17. Current participation in any other interventional clinical study within 30 days before the first administration of the investigational product or at any time during the study
18. Patients known or suspected of not being able to comply with this trial protocol
19. Patients of childbearing potential not willing to use adequate contraception during study and 3 months after last dose of therapy
20. Breast feeding women or women with a positive pregnancy test at Screening visit

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission (CR) and CR with incomplete blood count recovery (CRi) | 2 months
  Efficacy assessments

SECONDARY OUTCOMES:
CR and CRi in a pre-defined subgroup analysis in patients with complex karyotype | 2 months
  Efficacy assessments
CR and rate of combined CR/CRi and CR with negativity for minimal residual disease (CRMRD-) | 2 months
  Efficacy assessments
Duration of response (DOR) | 4 years
  Efficacy assessments
Event-free survival (EFS) | 4 years
  Efficacy assessments
Overall survival (OS) | 4 years
  Efficacy assessments
30-day and 60-day mortality | 30 and 60 days
  Safety assessments
Incidence and intensity of adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) version v4.0 | 12 months
  Safety assessments
Assessment of Quality of life by the EORTC Quality of Life Core Questionnaire (QLQ-C30) | 4 years
  Quality of life

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Kliniken Essen-Süd, Evang. Krankenhaus Essen-Werden gGmbH, Essen
  - Klinikum Oldenburg, Klinik für Innere Medizin II, Oldenburg
  - University Hospital Ulm, Ulm